CLINICAL TRIAL: NCT04493047
Title: mHealth for Pneumonia Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Maternal, Neonatal and Child Health Research Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16/136/109
Record Dates: First submitted 2020-04-17; First posted 2020-07-30 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2020-07

CONDITIONS: Pneumonia; Childhood Pneumonia; Infectious Disease; Acute Respiratory Infection
Keywords: childhood Pneumonia; Acute respiratory illness; Pakistan
MeSH Terms: conditions — Pneumonia; Communicable Diseases | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: The design of model will be based on the Replicating Effective Program (REP) framework of implementation. The first phase of REP is comprised of a systematic review (SR) on best mobile health based approaches for LHWs on management of childhood illness followed by formative research (FR). The study consists of the following three stages:
  * Pre-intervention phase
  * Intervention phase
  * Post-intervention phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Counselling on pneumonia prevention (Experimental): Recruited caregivers will be counselled by Lady health workers on pneumonia and its prevention via an audiovisual user friendly android based mobile application. Additionally, one text and one voice message will also be sent to the caregivers cell phones on the same subject.
  Interventions: Behavioral: Mobile health (mHealth) for pneumonia

INTERVENTIONS:
Behavioral: Mobile health (mHealth) for pneumonia — Audiovisual mobile based application will be used to counsel caregivers of children under five on pneumonia and its prevention. This will be coupled with text and voice message dissemination to the cell phones of caregivers.

SUMMARY:
In Pakistan, pneumonia and recurrent wheeze in children under five pose significant threats to children's health. Despite being preventable, more than 90,000 children die each year due to pneumonia in Pakistan, making it one of the top five countries in the world, with the highest pneumonia related childhood mortality. The predisposing factors which lead to these illnesses include lack of hygiene, lack of immunization, overcrowding, household air pollution, smoking, and poverty. Prompt recognition and timely initiation of treatment is imperative in children under five with pneumonia and recurrent wheeze and failure to do so can lead to complications and death. In children under five, among the causes of death due to these diseases, one is delayed care seeking. It has been identified that around 38% of deaths due to respiratory illnesses occur in households due to this delayed care seeking which is defined as delay in care sought for an illness outside home.

DETAILED DESCRIPTION:
In most of the low middle income countries, carer gender plays an important role in decisions to seek care. Although in majority of households, the primary caregivers of children under five are the mothers of those children, decisions with respect to care are often made by fathers or mothers in law which is a problem as they do not cater to the child in a timely manner either by not being there or being ignorant of basic management of the illness. Another contributing factor could be lack of time to take the child for healthcare as the mothers are usually occupied in their household chores and the fathers are busy working. And in rare cases where either the mother of a child dies at childbirth (500 per 100,000 live births) and when fathers are working away from home, it is the secondary caregiver who is responsible for care seeking of that child. Additionally, due to poverty, most caregivers cannot afford the cost of travel and secondary care for the child delaying care seeking until the child is severely ill. The inaccessibility of adequate healthcare within close proximity may delay care seeking. However a major contributing factor to this delay is impaired carer perception of the seriousness of the condition. The importance of caregivers' ability to recognize and seek appropriate care for their children is also one of the recommended key activities in the World Health Organization's (WHO)and UNICEF's Global Action Plan for the Control of Pneumonia and Diarrhea [11]. WHO and UNICEF have, therefore, emphasized the development of innovative, sustainable and cost-effective strategies/interventions to improve child health. It is important to devise a strategy whereby patients' symptoms are identified timely and immediate care given at their doorstep. Experimental studies provide the strongest evidence that illness perceptions can modify behaviors and care-seeking, and several studies have shown that interventions designed to change illness perceptions can improve health outcomes.

The inaccessibility of adequate healthcare within close proximity may delay care seeking. However a major contributing factor to this delay is impaired carer perception of the seriousness of the condition. Although well-proven life-saving tools are available to stop mortality due to preventable illnesses like pneumonia and recurrent wheeze, the existing health systems in Pakistan are passive. One of the most impact strategies can be timely healthcare seeking through community health workers who have been a powerful force to promote healthy behaviors and extend the reach to the health system by acting as a bridge between the community and the system. Community-based packaged interventions delivered through CHWs have been shown to improve care seeking for childhood illnesses. In Pakistan, these CHWs are referred to as Lady Health Workers (LHWs) enrolled under the National Program for Family Planning and Primary Healthcare. On average each LHW covers 100-150 households by making monthly visits and providing basic health services and education. These LHWs could, therefore, be a useful mode as evidence has shown that health interventions integrating (CHWs) can lead to positive behavior changes and lower morbidity and mortality rates, while moving services and information closer to the communities where they are actually needed.

Thus, our study will explore care-seeking for childhood pneumonia among caregivers of children under five through a qualitative approach and devise a Care Model to actively find cases through LHWs and promote appropriate care seeking behavior.

Primary Objective

• To determine the feasibility of using an android based mobile application by LHWs to educate caregivers of children under five on prevention of pneumonia in rural Islamabad.

ELIGIBILITY:
Inclusion criteria for LHWs:

• LHWs that have been nominated by the district health officer (DHO).

Inclusion criteria for under five pneumonia caregivers

* Caregivers of all children under five years.
* Caregivers residing in the study site.
* Caregivers who can understand Urdu.
* Caregivers who will consent to participate.
* Those caregivers who have mobile phones in their household.

Exclusion criteria for LHWs:

• LHWs not assigned the catchment area households for visits.

Exclusion criteria for under five pneumonia caregivers:

• Any household with a child under five having a chronic debilitating illness.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Number of caregivers with improved knowledge on under five pneumonia | 6 months
  A structured questionnaire will be used to interview the caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tabish Hazir, MBBS, FRCPCH, Principal Investigator — Maternal, Neonatal and Child Health Research Network
Locations (1):
- MNCHRN, Islamabad, Federal, Pakistan